CLINICAL TRIAL: NCT04270058
Title: Pregnancy Surveillance Program of Women and Infants Exposed to TEGSEDI During Pregnancy
Brief Title: TEGSEDI Pregnancy Surveillance Program
Status: Not yet recruiting | Type: Observational
Sponsor: Akcea Therapeutics (Industry)
Responsible Party: Sponsor
Other Study IDs: TEG4005; EUPAS41839 (Other: EU PAS)
Record Dates: First submitted 2020-02-07; First posted 2020-02-17 (Actual); Last update posted 2025-08-19 (Actual); Status verified 2025-08

CONDITIONS: Hereditary Transthyretin-mediated Amyloidosis With Polyneropathy; Pregnancy
Keywords: Hereditary transthyretin amyloidosis with polyneuropathy; Hereditary transthyretin amyloidosis; hATTR; hATTR-PN; Rare disease
MeSH Terms: conditions — Amyloidosis, Hereditary, Transthyretin-Related; Rare Diseases | interventions — Inotersen

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 21 Months
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Cohort 1: Cohort 1 will be pregnant patients who have been exposed to at least 1 dose of TEGSEDI within 25 weeks prior to conception or during pregnancy.
  Interventions: Drug: inotersen
- Cohort 2: Cohort 2 will be pregnant patients who have hATTR-PN, who were not exposed to TEGSEDI or have not received TEGSEDI within the previous 25 weeks prior to conception.

INTERVENTIONS:
Drug: inotersen — TEGSEDI injection, for subcutaneous use
  Groups: Cohort 1

SUMMARY:
This is a worldwide safety surveillance study of pregnancy outcomes in women with hATTR-PN who may have been exposed or were not exposed to TEGSEDI prior to or during the pregnancy and of pediatric outcomes up to 1 year of age.

ELIGIBILITY:
Inclusion Criteria:

TEGSEDI exposed patients (Cohort 1) meeting the following criteria will be eligible for study entry:

1. Pregnancies exposed to at least 1 dose of TEGSEDI within 25 weeks prior to conception or during pregnancy.
2. Able and willing to provide informed consent.

Unexposed patients (Cohort 2) meeting the following criteria will be eligible for study entry:

1. Have a diagnosis of hATTR-PN during pregnancy.
2. Have not been exposed to TEGSEDI within 25 weeks prior to conception or during pregnancy.
3. Able and willing to provide informed consent.

Exclusion Criteria:

None

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Gender Based: Yes
Study Population: There will be 2 cohorts:
  Cohort 1 will be pregnant patients who have been exposed to at least 1 dose of TEGSEDI within 25 weeks prior to conception or during pregnancy.
  Cohort 2 will be pregnant patients who have hATTR-PN, who were not exposed to TEGSEDI or have not received TEGSEDI within the previous 25 weeks prior to conception.
  The exposed cohort will include pregnant patients from any country where TEGSEDI is marketed and/or clinical trials, post-market studies and registries are being conducted or expanded access programs are available.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2025-12 (Estimated); Primary Completion 2030-11-15 (Estimated); Study Completion 2030-11-15 (Estimated)

PRIMARY OUTCOMES:
Frequency of Selected Pregnancy and Fetal/Neonatal Outcomes | 10 years or 12 months after the last live birth whichever is later
  Estimate the frequency of selected pregnancy and fetal/neonatal outcomes through 1 year of age in women who were exposed to at least 1 dose of TEGSEDI (Cohort 1) within 25 weeks prior to conception or during pregnancy, with the exposure window of interest for major congenital malformations being the first trimester, and in the unexposed cohort of pregnant women (Cohort 2) who have a diagnosis of hereditary transthyretin amyloidosis with polyneuropathy (hATTR-PN)
  * pregnancy outcomes include live births, spontaneous abortions, stillbirths, elective abortions, preterm birth
  * fetal/neonatal outcomes include major and minor congenital malformations, small for gestational age, failure to thrive, and postnatal development
Frequency of Selected Pregnancy Complications | 10 years or 12 months after the last live birth whichever is later
  Estimate the frequency of selected pregnancy complications in women who were exposed to TEGSEDI (Cohort 1) within 25 weeks prior to conception or during pregnancy and in the unexposed cohort of pregnant women (Cohort 2) who have a diagnosis of hATTR-PN